CLINICAL TRIAL: NCT00508924
Title: A Randomised, Open, Parallel-group, Multicentre Study to Examine the Safety and Effectiveness of Three Doses of Argatroban as Anticoagulant in Combination With Clopidogrel and Aspirin in Patients Undergoing Elective Percutaneous Coronary Intervention in Comparison With Unfractionated Heparin, Clopidogrel and Aspirin
Brief Title: Study on Safety and Effectiveness of Three Doses of Argatroban as Anticoagulant in Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARG-E04
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Angina, Unstable
Keywords: Argatroban; Direct thrombin inhibitor; Percutaneous coronary intervention; Activated clotting time; PCI; ACT
MeSH Terms: conditions — Coronary Artery Disease; Angina, Unstable | interventions — argatroban; Heparin

ARMS (4):
- ARG250 (Experimental)
  Interventions: Drug: Argatroban
- ARG300 (Experimental)
  Interventions: Drug: Argatroban
- ARG350 (Experimental)
  Interventions: Drug: Argatroban
- Heparin (Placebo Comparator)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Argatroban
  Arms: ARG250
Drug: Argatroban
  Arms: ARG300
Drug: Argatroban
  Arms: ARG350
Drug: Heparin
  Arms: Heparin

SUMMARY:
This is a phase II multi-centre study in 140 patients undergoing elective PCI to obtain the information on dose-response of argatroban in pharmacodynamic markers and to assess the anticoagulation, safety and efficacy of argatroban in reference to unfractionated heparin, in combination with dual antiplatelet therapy.

DETAILED DESCRIPTION:
This is a phase II multi-centre study in Europe in patients with stable coronary artery disease or troponin negative unstable angina undergoing elective PCI, to obtain the information on the safety and effects on various pharmacodynamic markers, of three doses of argatroban in combination with clopidogrel and aspirin, and to assess the results of argatroban and unfractionated heparin, both used in combination with clopidogrel and aspirin, on clinical outcomes, adequacy of anticoagulation, various pharmacodynamic markers (approximately 35 patients per group).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (women of child bearing potential must have a negative pregnancy test prior to entry into the study)
* Aged over 18 years
* Diagnosis of stable coronary artery disease (CAD) or unstable angina (troponin negative, i.e. within the normal range for the study site) with low to moderate anatomic risk and a requirement for elective percutaneous coronary angioplasty or stent insertion with an approved device in one or more de novo-treated or re-stenotic lesions in native vessels
* Signed written informed consent

Exclusion Criteria:

* Any condition which, in the investigator's opinion, contraindicates the use of argatroban, heparin or clopidogrel or endangers the patient if he/she participated in this study.
* Known cirrhosis, hepatitis, clinically significant hepatic disorder, or history of hepatic disorder. Hepatic disorder is defined as having levels of liver function tests (bilirubin, Aspartate Aminotransferase (Serum Glutamate Oxaloacetate Transaminase)(AST (SGOT)), Alanine Aminotransferase (Serum Glutamate Pyruvate Transaminase)(ALT (SGPT)) greater than 3.0 times above the upper limit of the normal range of local laboratory.
* Patients not currently taking aspirin
* Renal insufficiency, defined as serum creatinine greater than 2.0 mg/dL (greater than 177mmol/L)
* Platelets less than 125,000/ml
* If already taking any form of heparin prior to study enrolment, Activated Partial Thromboplastin Time(aPTT) equal or greater than 35 sec or ACT greater than 160 sec
* Use of low molecular heparin (LMWH) during 12 h prior to PCI
* If taking oral anticoagulant medication prior to study enrolment, International Normalised Ratio(INR) greater than 1.2
* Q wave MI with cardiogenic shock or thrombolytic therapy within 72 h of study dosing
* Use of Glycoprotein IIb / IIIa(GPIIb/IIIa) inhibitors within prior 3 weeks
* Documented coagulation disorder or bleeding diathesis
* Lumbar puncture within the past 2 weeks
* History of previous cerebral aneurysm, haemorrhagic stroke, or thrombotic stroke within the past 6 months
* Active, uncontrolled peptic ulcer disease or any gastrointestinal bleeding or genitourinary bleeding within 3 months prior to study enrolment
* Major surgery, serious trauma, puncture of non-compressible vessel, or biopsy of parenchymal organ within prior 2 months
* Planned staged procedure, planned rotational atherectomy, directional coronary atherectomy, brachytherapy, or thrombectomy catheters
* Planned surgical intervention other than study procedure within next 7 days
* Presence of greater than 50% stenosis of unprotected left main coronary artery
* Severe peripheral vascular disease, precluding femoral access
* History of vasculitis
* Uncontrolled hypertension defined as greater than 180/120 mmHg
* Pregnancy (exclusion by routine urine test)
* Lactating woman
* Woman of children bearing age who are or were not using accepted contraceptive methods
* Participation in other clinical trials of investigational products within 3 months prior to study enrolment
* Terminally ill patients with a life expectancy of < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-08; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma Europe
Locations (8):
- Aalst, Belgium
- Germany (7):
  - Bad Nauheim
  - Cologne
  - Dachau
  - Düren
  - Frankfurt
  - Halle
  - Mainz

REFERENCES:
- [Result] Rossig L, Genth-Zotz S, Rau M, Heyndrickx GR, Schneider T, Gulba DC, Desaga M, Buerke M, Harder S, Zeiher AM; ARG-E04 study group. Argatroban for elective percutaneous coronary intervention: the ARG-E04 multi-center study. Int J Cardiol. 2011 Apr 14;148(2):214-9. doi: 10.1016/j.ijcard.2010.02.044. Epub 2010 Mar 11. PMID 20226548

RESULTS

PARTICIPANT FLOW:
Groups:
- ARG250: 250μg/kg i.v. bolus of argatroban followed by infusion of 15μg/kg/min
  additional 150μg/kg i.v. boluses (maximum 2 additional) could be given in order to reach the target ACT level of 250 sec
- ARG300: 300μg/kg i.v. bolus followed by infusion of 20μg/kg/min
  additional 150μg/kg i.v. boluses (maximum 2 additional) could be given in order to reach the target ACT level of 250 sec
- ARG350: 350μg/kg i.v. bolus followed by infusion of 25μg/kg/min
  additional 150μg/kg i.v. boluses (maximum 2 additional) could be given in order to reach the target ACT level of 250 sec
- Heparin: 70-100 IU/kg i.v. bolus
  additional 2,000-5,000 IU boluses could be given in order to reach the target ACT level of 250 sec
Period: Overall Study
Arm/Group | ARG250 | ARG300 | ARG350 | Heparin
Started | 36 | 38 | 32 | 34
Completed | 36 | 38 | 31 | 33
Not Completed | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARG250 | ARG300 | ARG350 | Heparin | Total
Number analyzed (Participants) | 36 | 38 | 32 | 34 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (8.9) | 65.5 (9.5) | 68.3 (7.9) | 65.9 (9.8) | 65.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 5 | 33
  Male | 25 | 30 | 23 | 29 | 107

OUTCOME MEASURES:

1. Primary Outcome: Activated Clotting Time (ACT) Value After the First Dosing of Study Treatment.
Time Frame: 5 - 10 min after initial bolus
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | ARG250 | ARG300 | ARG350 | Heparin
Number analyzed (Participants) | 36 | 38 | 31 | 33
second | 301.0 [262.8 to 330.0] | 330.0 [270.0 to 365.0] | 354.0 [307.0 to 391.0] | 237.5 [198.0 to 284.0]

2. Primary Outcome: Composite and Each of Death, Myocardial Infarction, and Urgent Revascularisation at Day 30, and Major Bleeding Events During Hospital Stay.
Description: Composite end point (a): all cause death, myocardial infarction and urgent revascularization at Day30
  Composite end point (b): all cause death, myocardial infarction and urgent revascularization at Day30 as well as major bleeding events during hospital stay
Time Frame: 30 Days
Measure: Number; unit: participants
Arm/Group | ARG250 | ARG300 | ARG350 | Heparin
Number analyzed (Participants) | 36 | 38 | 31 | 33
participants
  Composite end point (a) | 1 | 0 | 1 | 1
  Composite end point (b) | 1 | 0 | 1 | 2
  All cause death | 0 | 0 | 0 | 0
  Myocardial infarction | 0 | 0 | 1 | 1
  Urgent revascularization | 1 | 0 | 1 | 0
  Major bleeding | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | ARG250 | ARG300 | ARG350 | Heparin
Serious Adverse Events (participants affected / at risk) | 4/36 | 5/38 | 7/32 | 4/34
Other Adverse Events (participants affected / at risk) | 22/36 | 25/38 | 23/32 | 27/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARG250 (N=36) | ARG300 (N=38) | ARG350 (N=32) | Heparin (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Artrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Groin infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basilar migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARG250 (N=36) | ARG300 (N=38) | ARG350 (N=32) | Heparin (N=34)
Angina pectoris (Cardiac disorders) | 2 | 3 | 4 | 4
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 4
Catheter site haematoma (General disorders) | 12 | 9 | 9 | 10
Catheter site haemorrhage (General disorders) | 3 | 0 | 3 | 2
Catheter site pain (General disorders) | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 2 | 1 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Cardiac enzymes increased (Investigations) | 3 | 1 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 1 | 3
Haemoglobin decreased (Investigations) | 1 | 1 | 2 | 3
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 3
Troponin T increased (Investigations) | 2 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 0
Syncope vasovagal (Nervous system disorders) | 3 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 4 | 2 | 5
Hypotension (Vascular disorders) | 3 | 2 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other